CLINICAL TRIAL: NCT01082367
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Multi-Center Study to Assess the Efficacy and Safety of Inhaled Tobramycin Nebuliser Solution (TOBI®) for the Treatment of Early Infections of P. Aeruginosa in Cystic Fibrosis Subjects Aged From 3 Months to Less Than 7 Years
Brief Title: Randomized, Controlled Study of CF Patients Between 3 Months and Less Than 7 Years
Acronym: EARLY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTBM100C2304; 2009-016590-15 (EudraCT Number)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Treatment of Early Pulmonary Infections With P. Aeruginosa in Cystic Fibrosis Patients
Keywords: Tobramycin Inhalation solution; Cystic fibrosis; Lung disease; anti-bacterial agents
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- TOBI (tobramycin inhaled solution)/Placebo (Experimental): Participants randomized to TOBI received the investigational treatment for 28 days twice daily (bi)d in the first treatment cycle. At the end of first treatment cycle, participants who were positive for P. aeruginosa entered the open label (OL) phase of the study and received TOBI for 28 days bid. Participants who were negative for P. aeruginosa at the end of first treatment cycle and agreed to participate in the cross-over treatment period received placebo for 28 days bid (second treatment cycle).
  Interventions: Drug: TOBI; Drug: Placebo
- Placebo/TOBI (Placebo Comparator): Participants randomized to placebo group received 0.9 % saline (NaCl) for 28 days bid in the first treatment cycle. At the end of first treatment cycle, participants who were positive for P. aeruginosa entered the OL phase of the study and received TOBI for 28 days bid. Participants who were negative for P. aeruginosa at the end of first treatment cycle and agreed to participate in the cross-over treatment period received TOBI for 28 days bid (second treatment cycle).
  Interventions: Drug: TOBI; Drug: Placebo

INTERVENTIONS:
Drug: TOBI — TOBI (tobramycin inhaled solution)
Drug: Placebo — Placebo

SUMMARY:
This study investigated the efficacy of inhaled TOBI treatment for early infections of P. aeruginosa in paediatric patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* Early lower respiratory tract infection with P. aeruginosa,

Exclusion Criteria:

* Known local or systemic hypersensitivity to aminoglycosides or inhaled antibiotics.
* Administration of loop diuretics within 7 days prior to study drug administration.
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Alexandria, Egypt
- France (2):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Dresden, Germany
- Greece (2):
  - Novartis Investigative Site, Pátrai, Greece
  - Novartis Investigative Site, Thessaloniki, GR
- Hungary (4):
  - Novartis Investigative Site, Debrecen, Hungary
  - Novartis Investigative Site, Kaposvár, Hungary
  - Novartis Investigative Site, Szeged, Hungary
  - Novartis Investigative Site, Debrecen
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Bucharest, Romania
- Russia (3):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Yaroslavl
- Novartis Investigative Site, Zurich, Switzerland, Switzerland

REFERENCES:
- [Derived] Ratjen F, Moeller A, McKinney ML, Asherova I, Alon N, Maykut R, Angyalosi G; EARLY study group. Eradication of early P. aeruginosa infection in children <7 years of age with cystic fibrosis: The early study. J Cyst Fibros. 2019 Jan;18(1):78-85. doi: 10.1016/j.jcf.2018.04.002. Epub 2018 Apr 21. PMID 29685813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized 1:1 to TOBI or placebo. After 1 treatment cycle, participants who were P.a positive entered an OL phase. Participants who were P.a negative entered cross-over treatment.
Pre-assignment Details: The cross-over was optional. At the end of the cross-over or OL phase, participants who were P.a positive terminated the study. P.a negative participants entered follow-up.
Groups:
- TOBI (Tobramycin Inhaled Solution)/Placebo: Participants randomized to TOBI received the investigational treatment for 28 days twice daily (bi)d in the first treatment cycle. At the end of first treatment cycle, participants who were positive for P. aeruginosa entered the open label (OL) phase of the study and received TOBI for 28 days bid. Participants who were negative for P. aeruginosa at the end of first treatment cycle and agreed to participate in the cross-over treatment period received placebo for 28 days bid (second treatment cycle). Eligible participants were followed-up for up to 12-months, having visits every 3 months. If participants were detected P. aeruginosa positive, they received 28-days of OL TOBI. Participants who remained P.aeruginosa positive after TOBI OL treatment discontinued the study. Participants who became P.aeruginosa negative after OL TOBI treatment remained in the study.
- Placebo/TOBI: Participants randomized to placebo group received 0.9 % saline (NaCl) for 28 days bid in the first treatment cycle. At the end of first treatment cycle, participants who were positive for P. aeruginosa entered the OL phase of the study and received TOBI for 28 days bid. Participants who were negative for P. aeruginosa at the end of first treatment cycle and agreed to participate in the cross-over treatment period received TOBI for 28 days bid (second treatment cycle). Eligible participants were followed-up for up to 12-months, having visits every 3 months. If participants were detected P. aeruginosa positive, they received 28-days of OL TOBI. Participants who remained P.aeruginosa positive after TOBI OL treatment discontinued the study. Participants who became P.aeruginosa negative after OL TOBI treatment remained in the study.
Period: Double-blind Period
Arm/Group | TOBI (Tobramycin Inhaled Solution)/Placebo | Placebo/TOBI
Started | 26 | 25
Stage 1:1st Treatment (tx) Cycle | 26 | 25 (1 participant discontinued after cycle 1 due to an SAE)
Stage 2:no tx | 0 | 0
Entered OL TOBI | 4 | 18
P.A-free,Day 29 w/ no Cross-over | 9 | 0
Stage 3: Cross-over (co) tx | 13 | 6
Stage 4:no tx for Patients Not in co | 0 | 0
Completed | 21 | 12
Not Completed | 5 | 13
Not completed — Administrative problems | 0 | 1
Not completed — Lack of Efficacy | 5 | 11
Not completed — Adverse Event | 0 | 1
Period: Follow-up (F-U) Period
Arm/Group | TOBI (Tobramycin Inhaled Solution)/Placebo | Placebo/TOBI
Started | 19 | 10
Treated in F-U | 5 | 5
Completed | 17 | 9
Not Completed | 2 | 1
Not completed — Administrative problems | 1 | 0
Not completed — Abnormal lab values | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TOBI (Tobramycin Inhaled Solution)/Placebo | Placebo/TOBI | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 2.9 (1.96) | 2.7 (1.93) | 2.8 (1.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants P Aeruginosa-free After Completion of the First Treatment Cycle
Description: Sputum/throat swab cultures were assessed.
Time Frame: Day 29
Population: Intent-to-treat (ITT): The ITT included all randomized participants who received at least dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | TOBI (Tobramycin Inhaled Solution)/Placebo | Placebo/TOBI
Number analyzed (Participants) | 26 | 25
Percentage of participants | 84.6 | 24.0
Statistical Analysis 1: Comparison: TOBI (Tobramycin Inhaled Solution)/Placebo vs Placebo/TOBI; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 21.55, 95% CI 2-sided [4.67 to 99.52]

2. Secondary Outcome: Percentage of Participants Free From P. Aeruginosa 28 Days After Termination of the Second Treatment Cycle
Description: Sputum/throat swab cultures were assessed.
Time Frame: Day 91
Population: Cross-over participants from the ITT population were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | TOBI (Tobramycin Inhaled Solution)/Placebo | Placebo/TOBI
Number analyzed (Participants) | 13 | 6
Percentage of participants | 92.3 | 83.3

3. Secondary Outcome: Percentage of Participants P Aeruginosa-free at Termination of the Double Blind Period
Description: Sputum/throat swab cultures were assessed.
Time Frame: Day 91
Population: Participants from the ITT population, who were tested for microbiology, were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | TOBI (Tobramycin Inhaled Solution)/Placebo | Placebo/TOBI
Number analyzed (Participants) | 25 | 22
Percentage of participants | 76.0 | 47.8

ADVERSE EVENTS:
Groups:
- DB TOBI: DB TOBI
- DB Placebo: DB Placebo
- OL TOBI (Core): OL TOBI (core)
- Off-treatment (Core): Off-treatment (core)
- OL TOBI (Follow-up): OL TOBI (follow-up)
- Off-treatment (Follow-up): Off-treatment (follow-up)
Arm/Group | DB TOBI | DB Placebo | OL TOBI (Core) | Off-treatment (Core) | OL TOBI (Follow-up) | Off-treatment (Follow-up)
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/38 | 0/22 | 2/50 | 0/10 | 4/29
Other Adverse Events (participants affected / at risk) | 12/32 | 18/38 | 10/22 | 13/50 | 2/10 | 23/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB TOBI (N=32) | DB Placebo (N=38) | OL TOBI (Core) (N=22) | Off-treatment (Core) (N=50) | OL TOBI (Follow-up) (N=10) | Off-treatment (Follow-up) (N=29)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB TOBI (N=32) | DB Placebo (N=38) | OL TOBI (Core) (N=22) | Off-treatment (Core) (N=50) | OL TOBI (Follow-up) (N=10) | Off-treatment (Follow-up) (N=29)
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 5
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Oral mucosal eruption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 3 | 2 | 5 | 0 | 10
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 4
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 5
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Perineal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Acinetobacter test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Aspergillus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Pseudomonas test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 2
Streptococcus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 4 | 3 | 1 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4 | 0 | 7
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.